CLINICAL TRIAL: NCT06282861
Title: The ANTES B+ Study: An Open-label, Pragmatic, Randomized, Controlled Trial of Triple Therapy Versus LABA-LAMA Combination to Improve Clinical Control in High Risk GOLD B Patients (B+)
Brief Title: ANTES B+ Clinical Trial
Acronym: ANTES B+
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Delays in the opening and activation of participating sites, and a low recruitment rate, with only 48 participants enrolled over the course of one year
Sponsor: Fundacio Privada Mon Clinic Barcelona (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANTES B+; 2023-507304-32 (EudraCT Number)
Record Dates: First submitted 2024-02-13; First posted 2024-02-28 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; ECOPD; eosinophil; Trelegy; Clinical Control
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol; Formoterol Fumarate; indacaterol; olodaterol; Salmeterol Xinafoate; Glycopyrrolate; Tiotropium Bromide; GSK573719

STUDY DESIGN:
Intervention Model Description: Phase IV, open-label, prospective, pragmatic, interventional, randomized (1:1), multicenter, controlled, 12-month follow-up trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trelegy (Experimental): Trelegy commercial product. 1 inhalation daily for 12 months
  Interventions: Drug: Trelegy Ellipta 100/62.5/25Mcg Inh 30D
- LABA-LAMA (Active Comparator): Any LABA-LAMA combination approved in Spain is accepted. To be used according to product specifications for 12 months.
  Interventions: Drug: Brimica; Drug: Duaklir; Drug: Ultibro; Drug: Ulunar; Drug: Xoterna; Drug: Anoro; Drug: Laventair; Drug: Spiolto Respimat; Drug: Yanimo; Drug: Foradil; Drug: Broncoral; Drug: Formoterol stada; Drug: Oxis; Drug: Formatris; Drug: Formoterol Aldo; Drug: Onbrez; Drug: Oslif; Drug: Hirobriz; Drug: Striverdi; Drug: Beglan; Drug: Betamican; Drug: Inaspir; Drug: Serevent; Drug: Soltel; Drug: Eklira; Drug: Bretaris; Drug: Seebri; Drug: Tovanor; Drug: Enurev; Drug: Spiriva; Drug: Tavulus; Drug: Sirkava; Drug: Braltus; Drug: Gregal; Drug: Incruse; Drug: Rolufta

INTERVENTIONS:
Drug: Trelegy Ellipta 100/62.5/25Mcg Inh 30D — Product to be used according to specifications. 1 inhalation daily for 12 months
  Other Names: LABA/LAMA/ICS
  Arms: Trelegy
Drug: Brimica — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Duaklir — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Ultibro — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Ulunar — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Xoterna — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Anoro — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Laventair — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Spiolto Respimat — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Yanimo — As per product specifications
  Other Names: LABA/LAMA
  Arms: LABA-LAMA
Drug: Foradil — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Broncoral — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Formoterol stada — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Oxis — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Formatris — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Formoterol Aldo — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Onbrez — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Oslif — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Hirobriz — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Striverdi — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Beglan — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Betamican — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Inaspir — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Serevent — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Soltel — As per product specifications
  Other Names: LABA
  Arms: LABA-LAMA
Drug: Eklira — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Bretaris — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Seebri — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Tovanor — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Enurev — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Spiriva — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Tavulus — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Sirkava — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Braltus — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Gregal — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Incruse — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA
Drug: Rolufta — As per product specifications
  Other Names: LAMA
  Arms: LABA-LAMA

SUMMARY:
Current guidelines recommend initial treatment with dual long-acting bronchodilator therapy (LABA-LAMA) in patients with Chronic Obstructive Pulmonary Disease (COPD) of group B (defined by CAT≥10 and none or 1 moderate exacerbation). However, the investigators hypothesize that there is a subgroup of B patients (B+) at a particularly high risk for poor clinical control, characterized by the following:

* 1 moderate exacerbation in the previous year
* CAT≥10 despite current treatment with LABA -LAMA
* Blood eosinophil levels of ≥150 cells/ml

the investigators further hypothesize that B+ patients could benefit from triple therapy treatment (LABA-LAMA + Inhaled Corticosteroids). Therefore, the main goal of this clinical trial is to compare the efficacy of Trelegy (triple therapy) in improving clinical control in GOLD B+ patients with chronic obstructive disease when compared to standard double therapy (LABA -LAMA).

The clinical control is a validated composite endpoint that includes two domains, the patient's stability, and the impact of the disease.

1028 patients will be randomly allocated to receive either the standard therapy or Trelegy and will be monitored by the investigators for 1 year in 2 on-site visits + 2 remote visits.

ELIGIBILITY:
Inclusion Criteria:

* Female or male
* 40-80 yrs. of age
* Current/former smokers ≥10 pack-year
* Diagnosis of COPD according to GOLD 2023 (post-bronchodilator(BD) FEV1/FVC<0.7 in the appropriate clinical context) with FEV1 post-BD 30-70% of the reference value
* B+ phenotype

  * CAT≥10 despite being on LABA-LAMA for ≥3 months, and
  * 1 moderate ECOPD in the previous year (treated with a short course of oral steroids and/or antibiotics), and
  * ≥150 blood Eos/ μL (as determined by a single Eos measurement in the previous 12 months available in the medical record of the patient)
* A signed and dated written informed consent prior to study participation.

Exclusion Criteria:

* GOLD E (≥2 moderate or 1 severe ECOPD in the previous year)
* ICS treatment (or oral steroid for whatever reason) during the last 8 weeks (10)
* ECOPD during the last 8 weeks
* Current diagnosis of asthma or documented history of asthma in the medical record of the patient according to the 2023 Global Initiative for Asthma (GINA) guidelines or other accepted guidelines
* Other concomitant respiratory disease (e.g., bronchiectasis, lung fibrosis, lung neoplasm)
* Use of domiciliary long-term oxygen therapy or non-invasive ventilation
* Alpha-1 antitrypsin deficiency
* Unstable or life-threatening cardiac disease, including:

  * Myocardial infarction or unstable angina in the last 6 months
  * Unstable or life-threatening cardiac arrhythmia requiring intervention in the last 3 months.
  * New York Heart Association (NYHA) Class IV Heart failure.
* Participation on Pulmonary Rehabilitation Program within 4 weeks prior to Screening or subjects who plan to enter the acute phase of a Pulmonary Rehabilitation Program during the study.
* Long term antibiotic therapy (antibiotics are allowed for the short-term treatment of an exacerbation or for short term treatment of other acute infections during the study).
* Systemic, oral, parenteral corticosteroids used for COPD and/or other diseases in the 8 weeks before entering in the study (oral/systemic corticosteroids may be used to treat COPD exacerbations during the study).
* Active neoplasm
* Life expectancy < 1 yr.
* Current participation in other RCTs (randomized clinical trial)
* Non-compliance: subjects at risk of non-compliance, or unable to comply with the study procedures.
* Any disease, disability, or geographic location that would limit compliance for scheduled visits.
* Known allergy to Trelegy® components (vilanterol, umeclidinium and/or fluticasone furoate) or inability to use the Ellipta® device.
* Women who are pregnant or lactating or are planning to become pregnant during the study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Clinical Control (CC) | 3,6,9 and 12 months
  Patient persistently controlled by CC at all study visits (a subject to be categorized as having clinical control they must meet the criteria at month 3, 6, 9 and 12).

SECONDARY OUTCOMES:
Clinical Important Deterioration (CID) | 3,6,9 and 12 months
  Patients persistently non deteriorated by CID-CAT at all study visits.(a subject to be categorized as having control by CID-CAT they must meet the criteria a month 3, 6, 9 and 12).
Patients persistently controlled | 3,6,9 and 12 months
  Patients persistently controlled (at all visits) throughout the study between the two study arms as per:
  * CC - Stability Domain
    1. General status since the last visit
    2. Exacerbations in the last 3 months
  * CC - Impact Domain
    1. Sputum color
    2. Rescue medication use
    3. Minutes walked per day
    4. Dyspnea (mMRC)
  * CID-CAT - Exacerbations
  * CID-CAT - (Patient reported outcomes)PROs
  * CID-CAT - Lung function
Time to deterioration | 3,6,9 and 12 months
  time to first event of not being CC or suffer CID-CAT
Time to no control event of CC - Stability Domain | 3,6,9 and 12 months
  Time to first no control event for CC - Stability Domain
Time to no control event of CC - Impact Domain | 3,6,9 and 12 months
  Time to first no control event for CC - Impact Domain
Time to deterioration event of CID-CAT Exacerbations | 3,6,9 and 12 months
  Time to deterioration event for CID-CAT Exacerbations
Time to deterioration event of CID-CAT Spirometry | 3,6,9 and 12 months
  Time to deterioration event for CID-CAT Spirometry
Exacerbation rate | 3,6,9 and 12 months
  To compare several Health status related endpoints between study arms including:
  d.To evaluate the mean and annual rate of:
  * Moderate exacerbations (ECOPD)
  * Severe ECOPD (hospitalized)
  * Moderate and Severe ECOPD
Time to first Exacerbation | 3,6,9 and 12 months
  To compare several Health status related endpoints between study arms including:
  e.To evaluate time to first ECOPD including:
  * Moderate ECOPD
  * Severe ECOPD (hospitalized)
  * Moderate or Severe ECOPD
Spirometry changes | 3,6,9 and 12 months
  To compare several Health status related endpoints between study arms including:
  f. To assess annual FEV1(Forced Expiratory volume) and FVC (forced vital capacity) changes (ml/year)
Independent predictors | 3,6,9 and 12 months
  Independent predictors with a potential negative impact on achieving the CC, each of its domains and each of its variables at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Àlvar Agustí, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No